CLINICAL TRIAL: NCT03140969
Title: An Open-label, Multiple Dose, Dose Escalation Study to Evaluate the Safety and Tolerability of QR-110 in Subjects With Leber's Congenital Amaurosis (LCA) Due to c.2991+1655A>G Mutation (p.Cys998X) in the CEP290 Gene
Brief Title: Study to Evaluate QR-110 in Leber's Congenital Amaurosis (LCA) Due to the c.2991+1655A>G Mutation (p.Cys998X) in the CEP290 Gene
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Collaborators: Sepul Bio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PQ-110-001; 2017-000813-22 (EudraCT Number)
Record Dates: First submitted 2017-05-01; First posted 2017-05-04 (Actual); Results first posted 2022-12-27 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Leber's Congenital Amaurosis
Keywords: CEP290; p.Cys998X; c.2991+1655A>G; RNA therapy; Antisense oligonucleotide; Leber's congenital amaurosis
MeSH Terms: conditions — Optic Atrophy, Hereditary, Leber; Meckel Syndrome, Type 4

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- QR-110 (Experimental): Administered every 3 months
  Interventions: Drug: QR-110

INTERVENTIONS:
Drug: QR-110 — RNA antisense oligonucleotide for intravitreal injection
  Other Names: Sepofarsen

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of QR-110 administered via intravitreal injection in subjects with LCA due to the CEP290 p.Cys998X mutation.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and tolerability of QR-110 administered via intravitreal injection in subjects with LCA due to the CEP290 p.Cys998X mutation. Subjects will receive QR-110 in one eye every 3 months, for a maximum of 4 doses. Up to 3 dose levels of QR-110 will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ≥ 6 years of age at Screening with a clinical diagnosis of LCA and a molecular diagnosis of homozygosity or compound heterozygosity for the CEP290 p.Cys998X mutation.
* Best-corrected visual acuity greater than or equal to light perception in both eyes and equal to or worse than LogMAR +1.0 (Snellen notation 20/200) in the worse eye and equal to or worse than LogMAR +0.7 (Snellen notation 20/100) in the contralateral eye.
* Detectable outer nuclear layer (ONL) in the area of the macula.
* An electroretinogram (ERG) result consistent with LCA.
* Clear ocular media and adequate pupillary dilation to permit good quality retinal imaging.

Exclusion Criteria:

* Syndromic disease.
* Pregnant or breast-feeding female.
* Any clinically significant cardiac disease or defect.
* One or more coagulation parameters outside of the normal range.
* Any ocular disease or condition that could compromise treatment safety, visual acuity or interfere with assessment of efficacy and safety.
* Prior receipt of intraocular surgery or intravitreal injection within 3 months prior to study start or planned intraocular surgery or procedure during the course of the study.
* Use of any investigational drug or device within 90 days or 5 half-lives of Day 1, whichever is longer, or plans to participate in another study of a drug or device during the PQ-110-001 study period.
* Any prior receipt of genetic therapy for LCA

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2019-10-02 (Actual); Study Completion 2019-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sepul Bio Chief Medical Officer, Study Director — Sepul Bio
Locations (3):
- United States (2):
  - University of Iowa, Iowa City, Iowa
  - Scheie Eye Institute, University of Pennsylvania, Philadelphia, Pennsylvania
- Ghent University Hospital and Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Russell SR, Drack AV, Cideciyan AV, Jacobson SG, Leroy BP, Van Cauwenbergh C, Ho AC, Dumitrescu AV, Han IC, Martin M, Pfeifer WL, Sohn EH, Walshire J, Garafalo AV, Krishnan AK, Powers CA, Sumaroka A, Roman AJ, Vanhonsebrouck E, Jones E, Nerinckx F, De Zaeytijd J, Collin RWJ, Hoyng C, Adamson P, Cheetham ME, Schwartz MR, den Hollander W, Asmus F, Platenburg G, Rodman D, Girach A. Intravitreal antisense oligonucleotide sepofarsen in Leber congenital amaurosis type 10: a phase 1b/2 trial. Nat Med. 2022 May;28(5):1014-1021. doi: 10.1038/s41591-022-01755-w. Epub 2022 Apr 4. PMID 35379979
- [Derived] Cideciyan AV, Jacobson SG, Ho AC, Garafalo AV, Roman AJ, Sumaroka A, Krishnan AK, Swider M, Schwartz MR, Girach A. Durable vision improvement after a single treatment with antisense oligonucleotide sepofarsen: a case report. Nat Med. 2021 May;27(5):785-789. doi: 10.1038/s41591-021-01297-7. Epub 2021 Apr 1. PMID 33795869
- [Derived] Miah KM, Hyde SC, Gill DR. Emerging gene therapies for cystic fibrosis. Expert Rev Respir Med. 2019 Aug;13(8):709-725. doi: 10.1080/17476348.2019.1634547. Epub 2019 Jun 27. PMID 31215818
- [Derived] Cideciyan AV, Jacobson SG, Drack AV, Ho AC, Charng J, Garafalo AV, Roman AJ, Sumaroka A, Han IC, Hochstedler MD, Pfeifer WL, Sohn EH, Taiel M, Schwartz MR, Biasutto P, Wit W, Cheetham ME, Adamson P, Rodman DM, Platenburg G, Tome MD, Balikova I, Nerinckx F, Zaeytijd J, Van Cauwenbergh C, Leroy BP, Russell SR. Effect of an intravitreal antisense oligonucleotide on vision in Leber congenital amaurosis due to a photoreceptor cilium defect. Nat Med. 2019 Feb;25(2):225-228. doi: 10.1038/s41591-018-0295-0. Epub 2018 Dec 17. PMID 30559420

RESULTS

PARTICIPANT FLOW:
Groups:
- QR-110 Low Dose: One 160 μg loading dose, followed by up to three 80 μg maintenance doses administered every 3 months, for up to 4 doses per subject.
- QR-110 Mid Dose: One 320 μg loading dose, followed by up to three 160 μg maintenance doses administered every 3 months, for up to 4 doses per subject.
- QR-110 High Dose: One 500 μg loading dose, followed by up to three 270 μg maintenance doses administered every 3 months, for up to 4 doses per subject.
Period: Overall Study
Arm/Group | QR-110 Low Dose | QR-110 Mid Dose | QR-110 High Dose
Started | 6 | 5 | 0
Completed | 6 | 5 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- QR-110 Low Dose: 160/80 μg Cohort
- QR-110 Mid Dose: 320/160 μg Cohort
- Total: Total of all reporting groups
Arm/Group | QR-110 Low Dose | QR-110 Mid Dose | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.7 (15.06) | 19.4 (6.88) | 21.7 (11.71)
Age, Customized [Count of Participants; unit: Participants]
  6 to < 18 years | 3 | 2 | 5
  18 to < 65 years | 3 | 3 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 4 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 5 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 5 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Frequency and Severity of Ocular Adverse Events in the Treatment and Contralateral Eyes
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | QR-110 Low Dose | QR-110 Mid Dose
Number analyzed (Participants) | 6 | 5
Participants | 6 | 5

2. Secondary Outcome: Frequency and Severity of Non-ocular Adverse Events
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | QR-110 Low Dose | QR-110 Mid Dose
Number analyzed (Participants) | 6 | 5
Participants | 6 | 5

3. Secondary Outcome: Change in Best-corrected Visual Acuity (BCVA)
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: logMAR
Groups:
- QR-110 Low Dose: 160/80 μg Cohort - Treated Eye
- QR-110 Mid Dose: 320/160 μg Cohort - Treated Eye
Arm/Group | QR-110 Low Dose | QR-110 Mid Dose
Number analyzed (Participants) | 6 | 5
logMAR
  Baseline (Absolute Values) | 2.597 (1.2738) | 2.990 (1.4153)
  Changes from Baseline - Visit 8 (M3) | -0.813 (1.0073) | -0.126 (0.2165)
  Changes from Baseline - Visit 13 (M6) | -0.903 (1.0189) | -0.122 (0.1801)
  Changes from Baseline - Visit 17 (M9) | -0.923 (1.0417) | 0.386 (0.9610)
  Changes from Baseline - Visit 21 (M12) | -0.927 (1.0492) | -0.106 (0.1545)

4. Secondary Outcome: Change in Full-field Stimulus Test (FST)
Description: Average Red Light Score
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: log cd/m2
Arm/Group | QR-110 Low Dose | QR-110 Mid Dose
Number analyzed (Participants) | 6 | 4
log cd/m2 | -0.7 (0.33) | -1.2 (0.82)

5. Secondary Outcome: Change in Full-field Stimulus Test (FST)
Description: Average Blue Light Score
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: log cd/m2
Arm/Group | QR-110 Low Dose | QR-110 Mid Dose
Number analyzed (Participants) | 6 | 4
log cd/m2 | -0.6 (0.76) | -0.9 (0.82)

ADVERSE EVENTS:
Time Frame: From the start of the study through to study completion (approx 1 year 11 months)
Arm/Group | QR-110 Low Dose | QR-110 Mid Dose
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 2/6 | 4/5
Other Adverse Events (participants affected / at risk) | 6/6 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QR-110 Low Dose (N=6) | QR-110 Mid Dose (N=5)
Cataract (Eye disorders) | 2 | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QR-110 Low Dose (N=6) | QR-110 Mid Dose (N=5)
Conjunctival haemorrhage (Eye disorders) | 4 | 4
Cataract (Eye disorders) | 3 | 4
Lenticular opacities (Eye disorders) | 1 | 3
Conjunctival hyperaemia (Eye disorders) | 1 | 2
Retinal degeneration (Eye disorders) | 0 | 2
Anterior chamber cell (Eye disorders) | 0 | 1
Cataract cortical (Eye disorders) | 1 | 0
Cataract subcapsular (Eye disorders) | 1 | 0
Conjunctival oedema (Eye disorders) | 0 | 1
Corneal lesion (Eye disorders) | 0 | 1
Cystoid macular oedema (Eye disorders) | 0 | 1
Diplopia (Eye disorders) | 0 | 1
Dry eye (Eye disorders) | 1 | 0
Eyelid cyst (Eye disorders) | 0 | 1
Eyelid oedema (Eye disorders) | 0 | 1
Hypotony of eye (Eye disorders) | 0 | 1
Injection site haemorrhage (Eye disorders) | 0 | 1
Lens disorder (Eye disorders) | 0 | 1
Metamorphopsia (Eye disorders) | 0 | 1
Post procedural complication (Eye disorders) | 0 | 1
Posterior capsule opacification (Eye disorders) | 0 | 1
Retinal cyst (Eye disorders) | 0 | 1
Vitreal cells (Eye disorders) | 0 | 1
Vitreous opacities (Eye disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution shall be free to publish, present, or use any Data and results arising out of its performance of the protocol. At least 30 days prior to submission for publication, institution shall submit to Sponsor for review and comment any proposed oral or written publication. Institution will consider any such comments in good faith but is under no obligation to incorporate Sponsor's suggestions. The review period for abstracts or poster presentations shall be 30 days.

DOCUMENTS (2):
  • Study Protocol (2018-08-08): https://cdn.clinicaltrials.gov/large-docs/69/NCT03140969/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-09): https://cdn.clinicaltrials.gov/large-docs/69/NCT03140969/SAP_001.pdf